CLINICAL TRIAL: NCT03228797
Title: A Comparison of Postoperative Outcomes Provided by a Continuous Preperitoneal Infusion Versus Ultrasound Guided Transversus Abdominis Plane Block for Abdominoplasty
Brief Title: A Comparison of Postoperative Outcomes Provided by a Continuous Preperitoneal Infusion Versus Ultrasound Guided Rectus Sheath Block for Midline Emergency Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Manar Mamdouh Fahmy Elsharkawi (Other Government)
Responsible Party: Sponsor-Investigator, Dr Manar Mamdouh Fahmy Elsharkawi, anaesthesiologist, Dubai Health Authority
Organization: Dubai Health Authority (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MRC-09/2014_07
Record Dates: First submitted 2017-07-06; First posted 2017-07-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Abdominal Pain
Keywords: pain
MeSH Terms: conditions — Abdominal Pain; Pain

STUDY DESIGN:
Intervention Model Description: comparative study between 3 groups using ropivacaine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (Active Comparator): ( 20 patients) will receive an ultrasound guided rectus sheath block by the end of the surgery using 15 ml ropivacaine 0.5% on either side.
  Interventions: Procedure: an ultrasound guided rectus sheath block
- Group II (Active Comparator): ( 20 patients) multiholed catheter will be inserted at the end of surgery and after the closure of the peritoneal layer, a10 ml bolus of ropivacaine 0.2% will be administered through the catheter and then connected to an elastomeric pump delivering a continuous fixed -rate of ropivacaine 5ml/h.
  Interventions: Procedure: multiholed catheter
- Group III (Active Comparator): ( 20 patients) a multiholed catheter will be inserted as in Group II and will receive also an ultrasound guided rectus sheath block as described for Group I.
  Interventions: Procedure: an ultrasound guided rectus sheath block &multiholed catheter

INTERVENTIONS:
Procedure: an ultrasound guided rectus sheath block
  Other Names: naropine 0.5%
  Arms: Group I
Procedure: multiholed catheter — gauge multiholed catheter will be inserted at the end of surgery and after the closure of the peritoneal layer at 3 to 5 cm away from the lower end of the surgical incision
  Other Names: naropine 0.2%
  Arms: Group II
Procedure: an ultrasound guided rectus sheath block &multiholed catheter — a multiholed catheter will be inserted as in Group II and will receive also an ultrasound guided rectus sheath block as described for Group I.
  Other Names: naropine 0.5% & naropine/ropivacaine 0.2%
  Arms: Group III

SUMMARY:
aim of this study is to compare the postoperative analgesia provided bya continuous preperitoneal infusion versus ultrasound guided rectus sheath block for midline emergency laparotomy.

anticoagulated patients

DETAILED DESCRIPTION:
Patients and Methods:

This randomized prospective study will be carried out after the approval of Rashid Hospital's Research Ethical Committee and patient's written informed consent.

Sixty adult patients , of both gender , 18-70 years old, ASA I-III who will be scheduled for emergency laparotomy with upper abdominal midline incision will be included in the study. Exclusion criteria will be patients with known allergic response or contraindications to paracetamol, parecoxib, morphine or ropivacaine and pregnant women

The enrolled patients will be randomly assigned to one of three groups:

Group I ( 20 patients) will receive an ultrasound guided rectus sheath block by the end of the surgery using 15 ml ropivacaine 0.5% on either side.

Group II ( 20 patients) for whom a 7.5 , 15 , 30 cm 19-gauge multiholed catheter will be inserted at the end of surgery and after the closure of the peritoneal layer at 3 to 5 cm away from the lower end of the surgical incision through an introducer peel-away needle. The length of the catheter will be established to guarantee homogenous distribution of the holes all along the length of the incision of the fascia. The catheter will be allocated above the peritoneum within the musculofascial layer and secured to the skin with an occlusive transparent dressing. A 10 ml bolus of ropivacaine 0.2% will be administered through the catheter and then connected to an elastomeric pump delivering a continuous fixed -rate of ropivacaine 10 ml/h.

Group III( 20 patients) a multiholed catheter will be inserted as in Group II and will receive also an ultrasound guided rectus sheath block as described for Group I.

No premedication will be administered. General anesthesia will be induced using target controlled intravenous infusion (TCI) using remifentanil (1-10 ng/ml effect concentration ) and propofol ( 1-10 mcg/ml effect concentration) titrated to Bi-spectral index (BIS) value between 40-60.Once anesthesia level will be reached , succinyl choline 1mg/kg intravenously will be given. After the airway will be secured , TCI will be adjusted to maintain BIS value between 40 to 60.An initial dose of 0.1 mg/kg intravenous cisatracurium will be administered and further doses will be given according to neuromuscular monitoring maintaining a train of four (TOF) value of zero.

Pre-incision , all patients will receive 15 mg/kg intravenous bolus and 40 mg intravenous parecoxib. 0.5 mg intravenous ketamine will be administered to avoid remifentanil's induced hyperalgesia.

All patients will be mechanically ventilated to maintain normocapnia throughout the procedure. Standard intraoperative monitoring will include electrocardiography, pulse oximetry , automatic non-invasive blood pressure , end tidal capnography , Bi-spectral index and train of four monitoring.

At the end of surgery and before extubation , patients who will be randomly assigned to Group I will receive an ultrasound-guided bilateral rectus sheath block using 15 ml of ropivacaine 0.5% on each side.

For patients who will be assigned to either Group II or Group III , a 7.5 , 15 or 30 cm 19-gauge multiholed catheter will be inserted by the operating surgeon at the end of surgery and after the closure of the peritoneal layer at 3 to 5 cm away from the lower end of the surgical incision through an introducer peel-away needle. The length of the catheter will be established to guarantee homogenous distribution of the holes all along the length of the incision of the fascia. The catheter will be allocated above the peritoneum within the musculofascial layer and secured to the skin with an occlusive transparent dressing. A 10 ml bolus of ropivacaine 0.2% will be administered through the catheter and then connected to an elastomeric pump delivering a continuous fixed -rate of ropivacaine 10 ml/h.

For patients who will be assigned to Group III will receive also an ultrasound-guided bilateral rectus sheath block using 15 ml of ropivacaine 0.5% on each side.

Then the patients will be extubated and shifted to Post-Anesthesia Care Unit (PACU) where they will be monitored for heart rate , blood pressure , oxygen saturation by pulse oximetry and pain score using visual analogue scale (VAS) both at rest and deep breathing . These data will be recorded every 15 minutes for the first hour.

After one hour , the patients will be discharged from PACU according to Modified Aldrete Scoring if they will reach a score of 9 or more. All patients will receive parecoxib 40 mg intravenously twice a day and paracetamol in a dose of 40 mg/kg intravenously in three divided doses regularly for 48 hours postoperatively.

In the postoperative period, all the patients will be evaluated for their hemodynamic variables ( heart rate , respiratory rate , arterial blood pressure and arterial oxygen saturation ) and postoperative analgesia using VAS at rest and with deep breathing at 2,4,8,12,18,24,36 and 48 hours postoperatively.

If the patient's VAS will reach 4 at any time in the 48 hours postoperatively, 0.1 mg/kg titrated intravenous morphine rescue analgesia will be administered and repeated if required to maintain VAS less than 4.

All patients will respond to a quality of life questionnaire (QR 40) at 24 and 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA-1 to ASA-3,emergency midline laparotomy

Exclusion Criteria:

* ASA-4 & above,allergic patients to the study's medications ,morbid obeses patients,patient refusal,age below 18yrs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
self reported pain intensity in the morning ,afternoon,evening, during activity over the past 2 days | 2 days
  each item is scored (0-10)0=no pain& 10= the worst

CONTACTS AND LOCATIONS:
Overall Officials: DR.HANY GREISS, consultant, Principal Investigator — DHA -Rashid hospital; DR.MANAR MAMADOUH, specialist, Principal Investigator — DHA -Rashid hospital; DR.MANSOUR NADHRI, consultant, Study Director — DHA -Rashid hospital; DR.OSAMA ALANI, senior specialist, Study Director — DHA -Rashid hospital

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03228797/Prot_SAP_000.pdf